CLINICAL TRIAL: NCT04985526
Title: The Significance of the Skin Microbiome in the Pathophysiology of Polymorphic Light Eruption
Brief Title: Skin Microbiome and Polymorphic Light Eruption
Acronym: PLE_microbio
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 33-196 ex 20/21
Record Dates: First submitted 2021-06-14; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Polymorphic Light Eruption
MeSH Terms: interventions — octenidine; 1-Propanol; 2-Propanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polymorphic light eruption patients (Experimental): PLE patients subjected to MED testing and photoprovocation
  Interventions: Other: Octeniderm (octenidine dihydrochloride, 1-propanol, 2- propanol)
- Healthy subjects (Other): Normal healthy subjects
  Interventions: Other: Octeniderm (octenidine dihydrochloride, 1-propanol, 2- propanol)

INTERVENTIONS:
Other: Octeniderm (octenidine dihydrochloride, 1-propanol, 2- propanol) — Administering Octeniderm (octenidine dihydrochloride, 1-propanol, 2- propanol) or 0,9% sodium chloride (as control agent) to the skin

SUMMARY:
Polymorphic light eruption (PLE) is the most common form among UV-inducible disorders with a prevalence of approximately 11-21% worldwide and a clear predisposition of women. Usually, within several hours after an intense UV exposure, most likely in spring or early summer, the formation of itchy skin lesions particularly at the upper arms and V-neck and neck is distinctive for PLE. It has been suggested that the development of a potential photo-induced antigen may initiate a delayed-type hypersensitivity reaction in PLE (causing the skin rash) and the microbiota of the skin may be involved. We thus hypothesized that eliminating the microbiota of the skin by disinfection may affect the formation of PLE. The concept of this study covers a combined interindividual and intraindividual half-body comparison of the skin reactions of disinfected and contralateral non-disinfected areas upon UV exposure in PLE patients and healthy subjects.

DETAILED DESCRIPTION:
UV-induced erythema and pigmentation is quantified by visual scoring and reflectance spectroscopy to determine the minimum erythema dose (MED) exploring the fields of an UV test ladder on the dorsal skin of the study subjects.

Investigations after determining the MED and consecutive photo provocations on 4 subsequent days (PLE group only) using solar simulated UV radiation with slight dose increments include a half-body site comparison of test areas located on the back of the subjects in a randomized, double blinded manner. The microbiota of a respective test area is removed by the disinfection with Octeniderm (octenidine dihydrochloride, 1-propanol, 2- propanol) whereas a control site remains non-disinfected (sham-treated with physiologic sodium chloride solution).

The PLE related symptoms are evaluated by a validated PLE score, which is composed as follows:

Affected skin area (AA) [range, 0-4] + skin infiltration (SI) [range, 0-4] + 0.4 pruritus (P) [range, 0-10]; ([total range 0-12].

As additional procedures, tape strips and skin swabs are taken immediately after UV exposures. The material is used for shotgun metagenomic sequencing of microbes and further analysis such as quantitative measures of antimicrobial peptides and urocanic acid levels. Furthermore, suction blisters are produced after MED testing and the last day of photo provocation [Time Frame: At day 3 and 6] to profile the inflammatory milieu of the skin by transcriptomics. The epidermal blister roof is used together with optional skin biopsies (PLE patients only) for various investigations, including H/E and immunohistochemical stainings and messenger ribonucleic acid (mRNA) analysis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PLE by typical patient history, typical histology of skin lesions and/or positive photo provocation test
* Healthy subjects

Exclusion Criteria:

* Presence or history of malignant skin tumors; dysplastic melanocytic nevus syndrome
* Photosensitive diseases such as porphyria, chronic actinic dermatitis, xeroderma
* pigmentosum, basal cell nevus syndrome
* Autoimmune disorders such as lupus erythematosus or dermatomyositis
* Antinuclear antibodies titer over 1:160 within 12 months prior study
* Systemic treatment of steroids and/or immunosuppressive drugs within 4 weeks prior the study start
* Systemic treatment of antibiotics within the last 6 weeks prior study
* Local treatment of anti-microbial treatment in the test field area within the last 6 weeks prior the study
* Systemic treatment of medications/drugs/ that could affect inflammatory responses within 2 weeks prior study
* Allergy on tape strips and/or adhesive material
* Psychiatric disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Quantification of PLE | 1 week
  determined by PLE score (range, 0-12) of photo provocation results (0 best, 12 worst)
Quantification of erythema score (range, 0-4) | 1 week
  determined by visual and spectroscopic erythema score
Quantification of pigmentation (range, 0-4) | 1 week
  determined by visual and spectroscopic erythema score

SECONDARY OUTCOMES:
Measurement of multiple cytokines (panel of 96 cytokines) | 1 week
  determined by transcriptomics
Assessment of multiple microbiomes of the skin (quantity and variety) | 1 week
  determined by metagenomics
Measurement of quantity and quality of multiple Antimicrobial peptides (AMP) | 1 week
  determined by proteomics
Measurement of concentration of cis/trans-urocanic acid | 1 week
  determined by high pressure liquid chromotography (HPLC)
Quantification of cellular skin infiltration (T cells, granulocytes and macrophages) | 1 week
  determined by hematoxylin and eosin (H/E) and immunohistochemical stainings

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wolf, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Department of Dermatology, Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided